CLINICAL TRIAL: NCT03226301
Title: A Prospective, Multicenter, Phase-II Trial of Ibrutinib Plus Venetoclax in Patients With Creatinine Clearance >= 30 ml/Min Who Have Relapsed or Refractory Chronic Lymphocytic Leukemia (RR-CLL) With or Without TP53 Aberrations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Nordic CLL Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HO141 CLL / VIsion trial
Record Dates: First submitted 2017-05-15; First posted 2017-07-21 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Chronic Lymphocytic Leukemia in Relapse; Chronic Lymphocytic Leukemia in Remission
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Intervention Model Description: All patients receive ibrutinib + venetoclax (with delayed start and ramp up of venetoclax from cycle 3) for the 15 cycles. Patients not achieving MRD negativity after cycle 12 (PB) AND/OR cycle 15 (PB+BM) continue on ibrutinib maintenance (non-randomized group). Patients achieving MRD negativity after cycle 12 (PB) AND cycle 15 (PB+BM) are randomized 1:2 between ibrutinib maintenance (arm A) and stopping treatment (observation, arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibrutinib until progression/relapse (Experimental): All patients receive ibrutinib + venetoclax (with delayed start and ramp up of venetoclax from cycle 3) for the 15 cycles.
  MRDpositive patients (PB and BM) will continue on Ibrutinib maintenance (non-randomized group) until progression/relapse
  Interventions: Drug: Ibrutinib + Venetoclax 15 cycles; Drug: Ibrutinib until progression/relapse
- Arm A (Experimental): All patients receive ibrutinib + venetoclax (with delayed start and ramp up of venetoclax from cycle 3) for the 15 cycles.
  MRD negative patients (PB and BM) will be randomized to Arm A or Arm B. Arm A: Ibrutinib until progression/relapse (Continuous ibrutinib treatment until toxicity or progression)
  Interventions: Drug: Ibrutinib + Venetoclax 15 cycles; Drug: Ibrutinib until progression/relapse
- Arm B (Experimental): All patients receive ibrutinib + venetoclax (with delayed start and ramp up of venetoclax from cycle 3) for the 15 cycles.
  MRD negative patients (PB and BM) will be randomized to Arm A or Arm B. Arm B: Observation until event.
  Patients randomized to Arm B will get reinitiation of therapy during the observation period in case of:
  * progression according to IWCLL criteria or
  * MRD≥10-3 (PB) and at least one month later MRD ≥10-2 (PB).
  Treatment reinitiation will consist of ibrutinib and venetoclax (with ramp up of venetoclax from cycle 1) for 12 cycles
  Interventions: Drug: Ibrutinib + Venetoclax 15 cycles; Drug: Possible reinitiation treatment: Ibrutinib + Venetoclax 12 cycles

INTERVENTIONS:
Drug: Ibrutinib + Venetoclax 15 cycles — Cycle 1 + 2: 420 mg ibrutinib, day 1-28 | Cycle 3: 420 mg ibrutinib, day 1-28 | 20 mg venetoclax, day 1-7 | 50 mg venetoclax, day 8-14 | 100 mg venetoclax, day 15-21 | 200 mg venetoclax, day 22-28 | Cycle 4-15: 420 mg ibrutinib, day 1-28 + 400mg venetoclax, day 1-28
Drug: Ibrutinib until progression/relapse — 420mg ibrutinib daily until progression/relapse
  Arms: Arm A; Ibrutinib until progression/relapse
Drug: Possible reinitiation treatment: Ibrutinib + Venetoclax 12 cycles — Cycle 1: 420 mg ibrutinib | 20 mg venetoclax, day 1-7 | 50 mg venetoclax, day 8-14 | 100 mg venetoclax, day 15-21 | 200 mg venetoclax, day 22-28 | cycles 2-12: 420 mg ibrutinib, day 1-28 + 400 mg venetoclax, day 1-28
  Arms: Arm B

SUMMARY:
The aim of the current trial is to evaluate if combination treatment with venetoclax + ibrutinib in patients with relapsed or refractory chronic lymphocytic leukemia (RR CLL) can lead to MRD negativity, which may induce long lasting remissions for MRD-negative patients randomized to stopping treatment after 15 induction cycles.

ELIGIBILITY:
Inclusion Criteria:

* Documented CLL or SLL requiring treatment according to IWCLL criteria after either being refractory to first line therapy or relapse after initial therapy.

  * Age at least 18 years.
  * Adequate bone marrow function defined as:

    * Absolute neutrophil count (ANC) >0.75 x 109/L
    * Platelet count >30,000 /μL 30 x 109/L.
    * Hemoglobin >8.0 g/dL (5 mmol/L) Unless directly attributable to CLL infiltration of the bone marrow, proven by bone marrow biopsy
  * Creatinine clearance (CrCL) ≥ 30ml/min calculated according to the modified formula of Cockcroft and Gault or directly measured with 24hr urine collection.
  * Adequate liver function as indicated

    * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN)
    * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of nonhepatic origin)
    * Prothrombin time (PT)/International normal ratio (INR) <1.5 x ULN and PTT (activated partial thromboplastin time [aPTT]) <1.5 x ULN (unless abnormalities are related to coagulopathy or bleeding disorder).
  * Negative serological testing for hepatitis B (HBsAg negative and anti-HBc negative; patients positive for anti-HBc may be included if PCR for HBV DNA is negative and HBV-DNA PCR is performed every month until 12 months after last dose), negative testing for hepatitis C RNA within 42 days prior to registration.
  * WHO/ECOG performance status 0-3 (appendix C), stage 3 only if attributable to CLL.
  * Negative pregnancy test at study entry (for women of childbearing potential).
  * Male and female subjects of reproductive potential must agree to use both a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete abstinence , or sterilized partner) and a barrier method (e.g., condoms, cervical ring, sponge, etc.) during the period of therapy and for 90 days after the last dose of study drug.
  * Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements.
  * Written informed consent.

Exclusion Criteria:

* Any prior therapy with ibrutinib and/or venetoclax.
* Transformation of CLL (Richter's transformation).
* Patients with a history of confirmed progressive multifocal leukoencephalopathy (PML).
* Malignancies other than CLL currently requiring systemic therapies or not being treated in curative intention before or showing signs of progression after curative treatment.
* Known allergy to xanthine oxidase inhibitors and/or rasburicase.
* Known bleeding disorders (e.g., von Willebrand's disease or hemophilia).
* Uncontrolled or active infection.
* Patients requiring treatment with a strong cytochrome P450 (CYP) 3A inhibitor (see appendix K). or anticoagulant therapy with warfarin or phenoprocoumon or other vitamin K antagonists. Please note: Patients being treated with NOACs can be included, but must be properly informed about the potential risk of bleeding under treatment with ibrutinib.
* History of stroke or intracranial hemorrhage within 6 months prior to registration.
* Major surgery within 28 days prior to registration.
* Use of investigational agents which might interfere with the study drug within 28 days prior to registration.
* Vaccination with live vaccines within 28 days prior to registration
* Steroid therapy within 7 days prior to registration, with the exception of inhaled steroids for asthma, topical steroids, steroids up to 25 mg of prednisolone daily to control autoimmune phenomenon's, or replacement/stress corticosteroids.
* Pregnant women and nursing mothers.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2017-06-23 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2026-06-21 (Estimated)

PRIMARY OUTCOMES:
Number of patients with progression free survival 27 months after starting treatment | 27 months after last patient in trial
  arm B of the study

SECONDARY OUTCOMES:
Number of patients with MRD negativity 27 months after starting treatment | 27 months after last patient in trial
  all arms of the study
Number of patients with progression free survival | 7 years after last patient in
  all arms of the study
Number of patients reinitiating treatment | 7 years after last patient in
  arm B of the study
Number of patients with treatment failure after reinitiating treatment | 7 years after last patient in
  arm B of the study
Number of patients initiating new CLL treatment | 7 years after last patient in
  all arms of the study
Number of patients with MRD negativity 12 (peripheral blood) and 15 months (peripheral blood and bone marrow) after starting treatment | 15 months after last patient in trial
  all arms of the study
Number of patients alive | 7 years after last patient in
  all arms of the study
Number of patients with complete remission, partial remission and stable disease and the duration of remission for each group | 7 years after last patient in
  all arms of the study
Number and grading of adverse events, serious adverse events and adverse events of special interest (bleeding, atrial fibrillation and tumorlysis) | 7 years after last patient in
  all arms of the study
Number of patients with improved quality of life (by EORTC QLQ-C30 and QLQ-CLL16 questionnaires) | 51 months after last patient in trial
  all arms of the study

CONTACTS AND LOCATIONS:
Locations (49):
- Belgium (5):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Brugge-AZBRUGGE, Bruges
  - BE-Bruxelles-STLUC, Brussels
  - BE-Haine-Saint-Paul-JOLIMONT, Haine-Saint-Paul
  - BE-Leuven-UZLEUVEN, Leuven
- Denmark (6):
  - DK-Aalborg-AALBORGUH, Aalborg
  - DK-Copenhagen-RIGSHOSPITALET, Copenhagen
  - DK-Herlev-HERLEV, Herlev
  - DK-Holstebro-HOLSTEBRO, Holstebro
  - DK-Odense-OUH, Odense
  - DK-Roskilde-ROSKILDE, Roskilde
- Finland (5):
  - FI-Helsinki-HUS, Helsinki
  - FI-Jyvaskyla-KSSHP, Jyväskylä
  - FI-Kuopio-KYS, Kuopio
  - FI-Tampere-TAYS, Tampere
  - FI-Turku-TYKS, Turku
- Netherlands (26):
  - NL-Alkmaar-NWZ, Alkmaar
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-AVL, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Enschede-MST, Enschede
  - NL-Gouda-GROENEHART, Gouda
  - NL-Groningen-UMCG, Groningen
  - NL-Heerlen-ATRIUMMC, Heerlen
  - NL-Helmond-ELKERLIEK, Helmond
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Rotterdam-MAASSTADZIEKENHUIS, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Sneek-ANTONIUSSNEEK, Sneek
  - NL-Den Haag-HAGA, The Hague
  - NL-Tilburg-ETZ, Tilburg
  - NL-Uden-BERNHOVEN, Uden
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zaandam-ZAANSMC, Zaandam
  - NL-Zwolle-ISALA, Zwolle
- Norway (2):
  - NO-Lørenskog-AKERSHUS, Lørenskog
  - NO-Trondheim-STOLAV, Trondheim
- Sweden (5):
  - SE-Boras-SASBORAS, Borås
  - SE-Linköping-REGIONOSTERGOTLAND, Linköping
  - SE-Luleå-SUNDERBY, Luleå
  - SE-Lund-SUH, Lund
  - SE-Uppsala-UPPSALAUH, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niemann CU, Dubois J, Nasserinejad K, da Cunha-Bang C, Kersting S, Enggaard L, Veldhuis GJ, Mous R, Mellink CHM, van der Kevie-Kersemaekers AF, Dobber JA, Poulsen CB, Razawy W, Hollestein R, Frederiksen H, Janssens A, Schjodt I, Dompeling EC, Ranti J, Brieghel C, Mattsson M, Bellido M, Tran HTT, Kater AP, Levin MD. Long-term follow-up of MRD-guided ibrutinib plus venetoclax in relapsed CLL: phase 2 VISION/HO141 trial. Blood Adv. 2025 Aug 12;9(15):3665-3675. doi: 10.1182/bloodadvances.2024015180. PMID 40249856
- [Derived] Kater AP, Levin MD, Dubois J, Kersting S, Enggaard L, Veldhuis GJ, Mous R, Mellink CHM, van der Kevie-Kersemaekers AF, Dobber JA, Poulsen CB, Frederiksen H, Janssens A, Schjodt I, Dompeling EC, Ranti J, Brieghel C, Mattsson M, Bellido M, Tran HTT, Nasserinejad K, Niemann CU. Minimal residual disease-guided stop and start of venetoclax plus ibrutinib for patients with relapsed or refractory chronic lymphocytic leukaemia (HOVON141/VISION): primary analysis of an open-label, randomised, phase 2 trial. Lancet Oncol. 2022 Jun;23(6):818-828. doi: 10.1016/S1470-2045(22)00220-0. PMID 35654052
- [Derived] Levin MD, Kater AP, Mattsson M, Kersting S, Ranti J, Thi Tuyet Tran H, Nasserinejad K, Niemann CU. Protocol description of the HOVON 141/VISION trial: a prospective, multicentre, randomised phase II trial of ibrutinib plus venetoclax in patients with creatinine clearance >/=30 mL/min who have relapsed or refractory chronic lymphocytic leukaemia (RR-CLL) with or without TP53 aberrations. BMJ Open. 2020 Oct 15;10(10):e039168. doi: 10.1136/bmjopen-2020-039168. PMID 33060089
- See also: Related Info — http://www.hovon.nl